CLINICAL TRIAL: NCT05173545
Title: Clinical Pharmacokinetics of Mitoxantrone Hydrochloride Liposome Injection in Recurrent/Refractory Lymphoma Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLM60-PK
Record Dates: First submitted 2019-07-31; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-11

CONDITIONS: Recurrent/Refractory Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mitoxantrone Hydrochloride Liposome Injection（12 mg/m2） (Experimental): itoxantrone Hydrochloride Liposome Injection（12 mg/m2）
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection
- Mitoxantrone Hydrochloride Liposome Injection（16 mg/m2） (Experimental): itoxantrone Hydrochloride Liposome Injection（16 mg/m2）
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection
- Mitoxantrone Hydrochloride Liposome Injection（20mg/m2） (Experimental): itoxantrone Hydrochloride Liposome Injection（20 mg/m2）
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome Injection — Every 28 days is a administration cycle, a total of 4 cycles.Until the subject's PD or intolerable or withdrawal (whichever occurs first).
  5% Glucose Injection drugs dissolved in 250 ml, intravenous drip for 60 minutes.

SUMMARY:
This is a single-center, open, randomized parallel group design study to investigate the pharmacokinetic characteristics of Mitoxantrone Hydrochloride liposome injection in the treatment of relapsed/refractory lymphoma after the first administration, and the safety and efficacy.

DETAILED DESCRIPTION:
The study was divided into three dosage groups: 12 mg/m2, 16 mg/m2 and 20 mg/m2,and three dosage groups were randomly divided into parallel groups.Every 28 days is a administration cycle, a total of 4 cycles.Until the subject's PD or intolerable or withdrawal (whichever occurs first).

In the study before administration of the first cycle to cycle second will set up 16 blood points,to calculate the pharmacokinetic parameters of total mitoxantrone and free mitoxantrone after the first administration.

ELIGIBILITY:
Inclusion criteria

Subjects must satisfy all the following conditions before enrollment:

1. Fully understand the clinical trail and sign the Informed Consent Form (ICF).
2. Ages range from 18 to 70 years (including 18 and 70 years), men and women are not limited.
3. Histopathologically and/or cytologically diagnosed relapsed/refractory lymphoma patients must undergo at least a first-line standard treatment for relapse or no remission and no better choice for advanced patients.
4. ECOG≤2.
5. The estimated survival time was at least 3 months.
6. The screening period of laboratory examination meet the following conditions, and 7 days before hematological evaluation during screening，subjects did not receive growth factor (long-acting granulocyte colony-stimulating factor needs 2 weeks interval), platelet or granulocyte transfusion:

   1. WBC≥3.5×109/L
   2. ANC≥1.5×109/L
   3. PLT≥75×109/L
   4. Hb≥90 g/L
   5. TBil≤1.5×ULN,If elevated bilirubin is caused by lymphoma invading the liver, the total bilirubin is allowed to be less than 3 x ULN.
   6. ALT/AST≤2.5×ULN，If the elevation is caused by lymphoma invading the liver, allow it to be less than 5 x ULN.
7. The toxicity of previous antineoplastic treatments was restored to ≤ 1 (except hair loss and pigmentation).
8. Female subjects were HCG negative in urine or blood (excluding menopause and hysterectomy)，men and women of childbearing age of the subjects take effective contraception during the experiment and 30 days of the end of last treatment.
9. Ability to visit on time and follow the procedures, limitations and requirements of the scheme.

Exclusion criteria

Subjects consistent with any one of the following conditions:

1. Subjects are consistent with one of the following conditions in the previous anti-tumor treatment history:

   1. Those receiving Mitoxantrone or Liposome-entrapped Mitoxantrone previously.
   2. Those receiving treatment of Adriamycin or other anthracyclines previously, with the total cumulative dose of > 360 mg/m2 (when converted to 1 mg Adriamycin, other anthracyclines shall be equivalent to 2 mg Epirubicin or 2 mg Pirarubicin or 2 mg Daunorubicin or 0.5 mg Idarubicin);
   3. Those receiving anti-tumor treatment (including chemotherapy, radiotherapy, hormone therapy or administration of TCM with anti-tumor activity) within 4 weeks prior to the first use of the study drug) or taking part in other clinical trials and accept medication in clinical trials;
   4. Those who have not yet fully recovered from previous surgical or invasive procedures.
2. Those with other malignant tumors previously or currently (except the non-melanoma skin basal cell carcinoma under effective control, breast/cervical carcinoma in situ, and other malignant tumors not treated but under effective control in the past five years).
3. Subjects with known or existing primary or metastatic central nervous system lymphoma or active brain metastasis
4. Cardiac dysfunction

   1. Male: QTc>450 ms, female: QTc>470 ms when ECG examination in the Research Center during the screening period;
   2. Clinically significant arrhythmias, including but not limited to complete left bundle branch block, Degree II atrioventricular block and PR interval > 250 ms;
   3. Any risk factor that might increase the QTc interval, e.g. hypokalaemia, inherited long-QT syndrome, with current administration of the drug for prolonging the QT interval or discontinuance for less than 15 days;
   4. Congestive heart failure of ≥Grade 2 in the New York Heart Association;
   5. Cardiac ejection fraction less than 50% or less than the lower limit of laboratory examination vale range of Research Center;
   6. Within six months prior to recruitment occurred myocardial infarction, unstable angina, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, clinical history of severe pericardial disease, or electrocardiographic evidence of acute ischemia or abnormal active conduction system.
5. Subjects with known history of immediate or delayed hypersensitivity to the similar drug and excipient of the study drug.
6. Hepatitis B and hepatitis C active infection (HBsAg positive and HBsDNA more than 1000 copies / mL; HCV RNA more than 1000 copies / mL).
7. Human immunodeficiency virus (HIV) infection.
8. Uncontrollable systemic diseases (such as uncontrollable hypertension, diabetes, etc.).
9. Pregnant or lactating women.
10. Investigator believe that subjects have any conditions that are not suitable for participating in the experiment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic indexes, Cmax Maximum concentration (Cmax) | Up to 28 days
  aximum concentration (Cmax) of Mitoxantrone Hydrochloride Liposome
Pharmacokinetic indexes, Tmax | Up to 28 days
  Time to Cmax (Tmax) of Mitoxantrone Hydrochloride Liposome
Pharmacokinetic indexes, Maximum concentration (Cmax,u) | Up to 28 days
  Maximum concentration (Cmax,u) of Mitoxantrone Hydrochloride Liposome

SECONDARY OUTCOMES:
progression-free survival(PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first（assessed up to 100 months）
  progression-free survival(PFS) of Mitoxantrone Hydrochloride Liposome

OTHER OUTCOMES:
Number of participants with Adverse Events (AEs) | From the initiation of the first dose to 28 days after the last dose
  Adverse Events will be coded using Medical Dictionary for Regulatory Activities (MedDRA). An AE is any untoward medical occurrence in a patient or clinical study participant temporally associated with the use of study investigational product (IP), whether or not considered related to the study IP. "Adverse event" means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related

CONTACTS AND LOCATIONS:
Overall Officials: Yunhong Huang, Master, Study Director — Cancer Hospital of Guizhou Province
Locations (1):
- Guizhou Cancer Hospita, Guiyang, Guizhou, China